CLINICAL TRIAL: NCT04332445
Title: Dermatological Assessment of Primary Dermal Irritability Accumulated, Sensitization, Photoallergy and Phototoxicity.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herbarium Laboratorio Botanico Ltda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HB032-19
Record Dates: First submitted 2020-03-27; First posted 2020-04-02 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Sensitivity, Contact
MeSH Terms: conditions — Dermatitis, Contact

STUDY DESIGN:
Intervention Model Description: Clinical trial, single-arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): subjects, 18-70 y, healthy
  Interventions: Other: Hyaluronic Acid Gel

INTERVENTIONS:
Other: Hyaluronic Acid Gel — Health care product - to be apllied on the subject's skin

SUMMARY:
This is a clinical study for health care product safety assessment. The research is going to conducted with 55 subjects, aged 18 to 70 years. The product is applied on the right and/or left participant back. After a wash out, the product is reapplied. Medical evaluation will be available throughout the study to assess possible adverse events. The main of the study is to observe the effects of the application of the product on the skin and prove the absence of irritability and/or allergy, photoallergy and phototoxicity.

DETAILED DESCRIPTION:
Subjects phototypes I to IV (according to Fitzpatrick classification). The products is applied over semi-occlusive dressings, remaing in contact with the skin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants;
* Non-injured skin in the test region;
* Agreement to adhere to the test procedures and requirements and to attend the institute on the day(s) and at the time(s) determined for the evaluations;
* Ability to consent to participation in the study;
* Phototype (Fitzpatrick): II and III;

Exclusion Criteria:

* Pregnant or breastfeeding women;
* Use of the following systemic drugs: antihistamines, non-hormonal anti-inflammatory drugs and corticoids;
* History of allergy to cosmetics, topical products or research product;
* Localized or widespread dermatological diseases or inflammatory dermatoses active and nerve damage in the test region;
* Personal or family pathological history of skin cancer;
* Use of topical or systemic photosensitizing medication;
* History of phototoxic, photoallergic reactions, dermatoses caused by light, atopy, pathologies aggravated or triggered by ultraviolet radiation;
* Photo-induced pathologies;
* Frequent exposure to the sun or tanning chambers;
* Participated in an allergenicity study in a period of less than 4 weeks from the start of the study;
* Skin marks in the experimental area that interfere with the evaluation of possible reactions;
* Active dermatoses;
* Forecast to take a bath in the sea, pool or sauna during the study;
* Participants who play water sports;
* Dermography;
* Use of the following topical or systemic drugs: immunosuppressants, antihistamines, non-hormonal anti-inflammatory drugs and corticoids up to 2 weeks prior to selection or, considering deposit corticoids, the interval shall be 1 month prior to selection;
* Treatment with acid vitamin A and/or its derivatives via oral or topical until

  1 month before the beginning of the study;
* Aesthetic and/or body dermatological treatment until 3 weeks before selection;
* Vaccination during the study or until 3 weeks before the study;
* Being participated in another clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-03 (Actual)

PRIMARY OUTCOMES:
Erythema degree or absence | 39 days
  Erythema evaluation according to International Contact Dermatitis Research Group

CONTACTS AND LOCATIONS:
Locations (1):
- Kosmoscience Ciência e Tecnologia Cosmética Ltda, Campinas, São Paulo, Brazil